CLINICAL TRIAL: NCT01620905
Title: Development of a Clinical Prediction Rule to Identify Patients With Neck Pain Likely to Benefit From Cervical Spine Manipulation and Exercise
Brief Title: Development of a Clinical Prediction Rulefor Neck Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Franklin Pierce University (Other); University of Colorado, Denver (Other); International Spine Pain Institute (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Associate Professor, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UNLVPT08072806
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Mechanical Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cervical spine manipulation (Experimental): Subjects received cervical spine manipulation
  Interventions: Procedure: Manipulation

INTERVENTIONS:
Procedure: Manipulation — Single level cervical spine joint manipulation

SUMMARY:
Cervical spine manipulation has been shown to be helpful for some patients with neck pain. This study sought to determine factors which were predictive of which patients with neck pain would benefit from manipulation.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 60 years
* primary report of neck pain with or without unilateral upper extremity symptoms
* baseline neck disability index score of 10 points (out of 50) or greater

Exclusion Criteria:

* any medical red flags suggesting that the etiology of symptoms might be nonmusculoskeletal
* diagnosis of cervical spinal stenosis (as identified in the patients' medical intake form)
* bilateral upper extremity symptoms
* evidence of central nervous system involvement
* history of whiplash injury within 6 weeks of the examination
* pending legal action regarding their neck pain
* 2 or more positive neurologic signs consistent with nerve root compression (changes in sensation, myotomal weakness, or decreased deep tendon reflexes)
* any history of cervical spine surgery, rheumatoid arthritis, osteoporosis, osteopenia, or ankylosing spondylitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Global Rating of Change Scale | 48 hours post intervention
  15 point likert scale rating perceived recovery

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 48 hours and 96 hours post intervention
  Average pain scores (0 - no pain to 10 - worst imaginable pain) taken for current rating, best in last 24 hours and worst in last 24 hours
Neck Disability Index | 48 hours and 96 hours post intervention
  10 item questionnaire measuring perceived disability (range 0 to 50)

CONTACTS AND LOCATIONS:
Locations (1):
- UNLV PT Department, Las Vegas, Nevada, United States